CLINICAL TRIAL: NCT04012515
Title: Production of a Device to Obtain Continuous Ambulatory Vestibular Assessment (CAVA) - Electrode Pad Appraisal Trial
Brief Title: CAVA: Electrode Pad Appraisal Trial
Acronym: CEPAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Dawson (Other)
Collaborators: University of East Anglia (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 261103 (25-02-19)
Record Dates: First submitted 2019-04-05; First posted 2019-07-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Tolerability of Wear of Electrode Pads
Keywords: ECG Electrodes; ambulatory monitoring; dermatology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAVA Electrode Pad Appraisal Trial Arm (Experimental): All trial participants are within this arm. All participants will wear the same selection of electrode pads and follow the same replacement schedules.
  Interventions: Device: Electrode Pads

INTERVENTIONS:
Device: Electrode Pads — Participants wear six electrode pads in total; three different types of pad, worn in the same positions on both sides of the face. The pads on the left-hand side of the face are replaced daily, and those on the right-hand side are replaced every other day. The pads do not administer a medical treatment or perform any other active function. The purpose of the intervention is to determine which combination of pad and replacement regime maximises the tolerability of wear over a 30-day period.

SUMMARY:
This trial requires healthy volunteers to wear a selection of CE marked electrodes for up to 30 days. The results from this trial will determine which electrodes should be used with the CAVA device, which is a medical device for monitoring dizziness.

DETAILED DESCRIPTION:
Dizziness is a common condition that is responsible for a significant degree of material morbidity and burden on our health service. There are multiple causes of dizziness, and these originate from pathologies affecting a large variety of different organ systems. Dizziness is usually episodic and short-lived, so when a patient presents to their health care provider, examination is often normal. As such, diagnosis is challenging and patients often experience significant delay in receiving a diagnosis. We have developed a device for monitoring dizziness and in 2018 we evaluated the device by undertaking a clinical trial involving healthy volunteers. Following the promising results from the first trial, we will conduct a second trial in 2019 on patients suffering from dizziness.

During the healthy volunteer trial, a minor issue was encountered relating to long-term daily wear of the device's electrode pads. Specifically, nine participants reported varying degrees of skin redness and inflammation beneath their electrode pads, mostly occurring after around two weeks of wear. The issue was self-limiting and resolved after a few days of non-wear. The team worked closely with a consultant dermatologist in order to monitor and manage this adverse event.

Since the issue was identified, the team has consulted with a number of people with relevant expertise in order to determine the causes of the issue and to find the most viable solution. Based on these discussions, we propose that the causes of this issue were due to a combination of wear duration, and/or repeated removal, and/or the specific type of electrode pad used. To confidently identify the cause of this issue and to evaluate a number of possible solutions, we intend to undertake a trial to evaluate the tolerability of alternative electrode pads and different patterns of wear.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over.
* Able to commit to 30 days of continuous wear of the electrode pads as per the study plan.
* Own a telephone.

Exclusion Criteria:

* Potential participants who have a history of dermatological disease, damage around the forehead, or fragile skin.
* Potential participants who have an allergy to plasters and/or medical adhesives.
* Potential participants who have taken part in a previous CAVA trial.
* Potential participants who are currently taking part in another trial.
* Unable to follow the testing protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
The maximum duration of comfortable wear of electrode pad | 1 month
  The maximum duration of comfortable wear will be calculated for each combination of electrode pad and wear regime, and the longest duration will determine the best electrode pad for use with the CAVA device.

CONTACTS AND LOCATIONS:
Overall Officials: John Phillips, Principal Investigator — Consultant ENT Surgeon
Locations (1):
- Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich, United Kingdom